CLINICAL TRIAL: NCT00843895
Title: Serotyping of Pneumococci
Brief Title: Multicenter Prospective Evaluation of the Incidence and Serotyes of Invasive Pneumoccocal Disease (IPD) Among Children Below 5 Years
Acronym: Pneumococci
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King Saud University (Other)
Responsible Party: King saud university, wyeth
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Screening
Other Study IDs: kingsadu
Record Dates: First submitted 2009-02-09; First posted 2009-02-13 (Estimated); Last update posted 2009-02-13 (Estimated); Status verified 2009-02

CONDITIONS: Pneumococcal Disease
Keywords: Laboratory based study; antibiotic susceptibilty; invasive strains
MeSH Terms: conditions — Pneumococcal Infections | interventions — Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Who Masked: Participant

INTERVENTIONS:
Biological: pneumococcal conjugate vaccine(prevenar) — to see the vaccine impact on pneumococcal diseases

SUMMARY:
The purpose of this study is to identify the S. pneumoniae serotypes strains and to determine antibiotic susceptibility.

ELIGIBILITY:
Inclusion Criteria:

* age less than 5 years

Exclusion Criteria:

* none

Ages: 3 Weeks to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2009-03; Primary Completion 2009-08 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Incidence and serotypes of invasive pneumococcal dis. | 6-8 months

SECONDARY OUTCOMES:
Antibiotic susceptibility | 6-8 months